CLINICAL TRIAL: NCT04103294
Title: Measuring Cowpea Consumption in Young Children and Pregnant Women in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: College of Health Sciences, University of Ghana, Legon (Unknown); Project Peanut Butter, Ghana (Unknown); Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201905103
Record Dates: First submitted 2019-06-12; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cowpea variety #1 (Experimental): 25g of cowpea daily for days 6-10, 50g of cowpea daily for days 11-15 and then 75g of cowpea daily for days 16-20. The pregnant women will receive 50g of cowpea daily for days 6-10, 100g of cowpea daily for days 11-15 and then 150g of cowpea daily for days 16-20
  Interventions: Dietary Supplement: cowpea variety #1
- cowpea variety #2 (Experimental): 25g of cowpea daily for days 6-10, 50g of cowpea daily for days 11-15 and then 75g of cowpea daily for days 16-20. The pregnant women will receive 50g of cowpea daily for days 6-10, 100g of cowpea daily for days 11-15 and then 150g of cowpea daily for days 16-20
  Interventions: Dietary Supplement: cowpea variety #2

INTERVENTIONS:
Dietary Supplement: cowpea variety #1 — two most popular varieties of cowpea currently consumed in the selected geographic area
  Arms: cowpea variety #1
Dietary Supplement: cowpea variety #2 — two most popular varieties of cowpea currently consumed in the selected geographic area
  Arms: cowpea variety #2

SUMMARY:
Current dietary assessment methods rely on self-report food intake such as food frequency questionnaires, 24-hr dietary recall, or diet diaries, and the prevalence of misreporting with these tools is estimated at 30-88%.A reliable and convenient way to measure the quantity of cowpea consumed by an individual. The hope is to identify a novel set of dietary biomarkers that will measure cowpea consumption, be free from participant recall bias, and serve to quantify legume intake. A total of 40 subjects, 20 children (9-21 months) and 20 pregnant women (>18 yr) will consume 3 distinct daily intake dosages of cooked cowpeas with the daily intake increased every 5 days. Urine samples will be collected 3 times during each 5-day period and blood spots will be collected during a washout period and at the end of the final 5-day period. Urine samples will undergo metabolite detection via ultra-performance liquid chromatography tandem mass spectrometry in positive and negative ion mode. Peaks are quantified using area-under-the-curve (AUC) and each metabolite is quantified in terms of its median-scaled relative abundance for the metabolite across the entire data set. A repeated measures 2-way ANOVA will be used to compare cowpea metabolite abundances over time and with respect to variation in an individual baseline levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between the ages of 9-21 months and pregnant women > 18 years of age and between 20-25 weeks of gestation.

Exclusion Criteria:

* Children with acute malnutrition, congenital abnormalities, chronic debilitation disease such as heart disease, cerebral palsy, or HIV infection. For the pregnant women they should also be free from acute malnutrition, without known complications such as gestational diabetes, pre-eclampsia, gestational diabetes, or hypertension

Min Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Metabolomic profiling of Urine and Plasma | 20 days
  The study will look at the levels of cowpea metabolite in urine after 20 days of consuming a diet with different cowpeas. Comparing the level of metabolites in urine at the end of study with the start after the participant consumes no cowpea for 5 days after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- College of Health Sciences, University of Ghana, Accra, Mion and Nanton District, Ghana